CLINICAL TRIAL: NCT04670861
Title: Innovative Use of Biodex Balance System to Improve Dynamic Stabilization and Function of Upper Quarter in Recreational Weightlifters: A Randomized Controlled Trial
Brief Title: Effectiveness of Upper Quarter Biodex Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Almaz Abdel-Aziem, Professor of Biomechanics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PT. REC.012.002982
Record Dates: First submitted 2020-12-10; First posted 2020-12-17 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Resistance Training
Keywords: Biodex; Balance; Functional test; weightlifters; upper quarter

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Upper extremity Biodex balance training program three times/week for eight weeks in addition to regular weightlifting training exercises
  Interventions: Procedure: Upper extremity Biodex balance training
- control group (Active Comparator): regular weightlifting training exercises
  Interventions: Procedure: Upper extremity Biodex balance training

INTERVENTIONS:
Procedure: Upper extremity Biodex balance training — The person assumes the prone plank posture with both hands poisoned in the area assigned for foot placement on the tilting balance platform. Using the four keypads, the person's left hand, left wrist, right hand and right wrist positions are entered into the system using the midline of the hand and the platform grid as reference points. The dot that appears on the position patient screen represents the person's segmental center of gravity.
  During each trial test, the person should shift his weight to move the cursor from the center along a target path and back as quickly and with a little deviation as possible. The same process is repeated for each of the targets. Target paths activate in a random order.

SUMMARY:
Strength, and proprioception training of upper body following injuries is commonly recommended. However, there are no previous studies investigated the effects of Biodex balance training on the strength, stability and function of the upper quarter. So, the purpose of this study will investigate the effect of Biodex balance training on improving the strength, dynamic stability and function of the upper quarter in young recreational weightlifters.

DETAILED DESCRIPTION:
Study design This is randomized controlled study. There are two groups classified randomly (group A & group B); group (A); will receive upper extremities biodex balance training. 3 times/week for 8 weeks and group B that receive no treatment just assessment pre and post. Both groups will receive their regular weightlifting training exercises 4times/week.

Procedures Testing procedures Data collection from the testing procedures in the pre and post interventional phase will take place over two days to avoid the impact of fatigue on the participants' physical performance. In the first day, descriptive data will be measured and recorded for each subject including age, height, weight, upper extremity dominance (defined as the hand reported to be preferred for ball throwing). This will be followed by the upper quarter Y- balance (UQ-YBT) and the Dynamic limits of stability (DLOS) using the Biodex balance system. In the second day, data will be collected from the 2-minutes 90° push-up test and the one-arm hop test. The order of days and testing procedures will be randomized for all participants.

Training procedure Total number of 24 training sessions will be scheduled to the participants in group A over a period of eight weeks (three sessions/week). The Rating of perceived exertion (RPE) or Modified Borg scale (MBS) was used to monitor and guide exercise intensity. The scale allowed participants to subjectively rate their level of exertion during training. It starts at number 0 where training is causing no breathing difficulty at all and progress through to number 10 where breathing difficulty is maximal. Training will start with the current level of balance of each participant at which he reports exertion level of ≥ 5 based on modified Borg scale and progressed towards the more difficult ones. The Biodex display screen will be connected to a computer screen that will be positioned at a level to allow visual feedback to the participants during training The transition from one level to the more difficult one will be based on composite score of > 95% at the present level. Each training session will consist of three minutes training and one-minute rest, repeated for a total of 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy recreational male weightlifters aged between 19 and 25 years

Exclusion Criteria:

* if they took any hormonal supplements, participated in professional bodybuilding or power lifting competition, had shoulder pain or history of surgery or musculoskeletal injuries and if they dropped out their gym workout for more than three weeks in the last six months.

Ages: 19 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — A fifty male weightlifters
Enrollment: 50 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Upper quarter Y-balance | 8weeks (pre/post)
  The YBT-UQ consists of a platform to which three wooden rulers are attached in the medial, inferolateral, and superolateral reach directions. Each of the posterior rulers is positioned 135ᵒ from the anterior one. The posterior rulers are separated by a 90ᵒ angle between them.
Biodex limits of stability | 8weeks (pre/post)
  Dynamic stabilization of the upper quarter assessment and training was provided using Biodex SD system (Biodex, Inc., Shirley, NY, USA) to measure the composite score of the limits of stability (LOS). The system has a moveable multiaxial circular balance platform which can provide up to 20° of surface tilt within a 360° range of motion. The BBS is reported to be valid and reliable for balance assessment and treatment

SECONDARY OUTCOMES:
Two minutes (2-min) 90° push-up | 8weeks (pre/post)
  The exercise was performed on a flat, stable surface, hands placed slightly wider than shoulder-width apart, and fingers pointed forward. The participant "begins" the push-up by bending the elbows and lowering the body as a single unit until the upper arms are at least parallel to the ground (90° push-up) and then return to the starting position by raising the entire body until full extension of the arms. The aim of this test is to perform the maximum number of repetitions in two minutes
One-arm hop | 8weeks (pre/post)
  The subjects were instructed to perform two sets of 10 standard 2-hand push-ups with 2-minute rest period in-between as warming up. This was followed by familiarization trials of the one arm hop test with the dominant and nondominant upper extremities. The subject first watched an instructional video depicting the one-arm hop test.